CLINICAL TRIAL: NCT05135897
Title: The Neurobiological Fundaments of Depression and Its Relief Through Neurostimulation Treatments
Acronym: FundECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 254425
Record Dates: First submitted 2021-10-08; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorder 1; Major Depressive Disorder; Healthy
MeSH Terms: conditions — Major Depressive Disorder 1; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients, depression, ECT: Patients in major depressive episode undergoing ECT
  Interventions: Device: Electroconvulsive therapy
- Patients, depression, TMS: Patients in major depressive episode undergoing TMS
  Interventions: Device: rTMS
- Healthy: Healthy controls who do not receive ECT nor TMS but otherwise the same assessments.

INTERVENTIONS:
Device: Electroconvulsive therapy — Treatment with Electroconvulsive therapy
  Groups: Patients, depression, ECT
Device: rTMS — repetitive Transcranial Magnetic Stimulation
  Groups: Patients, depression, TMS

SUMMARY:
The study will apply state of the art radiology through advanced magnetic resonance imaging (MRI) techniques to investigate structural and functional brain effects of electroconvulsive therapy (ECT) and repetitive transcranial magnetic stimulation (rTMS).

DETAILED DESCRIPTION:
As a multi-disciplinary collaboration, imaging findings will be correlated to psychiatric response parameters, neuropsychological functioning as well as neurochemical and genetic biomarkers that can elucidate the underlying mechanisms. The aim is to document both treatment effects and potential harmful effects of ECT and TMS

Sample, three groups:

ECT: n = 50 patients in a major depressive episode (bipolar and major depressive disorder) who have accepted treatment with ECT.

TMS: n = 50 patients in a major depressive episode (bipolar and major depressive disorder) who have accepted treatment with TMS.

HC: = 50 age and gender matched healthy volunteers not receiving ECT nor TMS.

Observation time: six months, with the time points as specified below. ECT is typically given three times weekly, but exceptions may occur. Hence, time points are specified as the number of ECT treatments given rather than an exact number of days which will vary.

Tp1: 2 hours before the first treatment session (day 1, baseline), Tp2: 2 hours after the first treatment session (day 1), Tp3: before the 7th ECT session and corresponding time point for TMS (~ day 15), Tp4: 1-2 weeks after last treatment session (~ day 30 - 50), Tp5: 6 months after treatment (~ day 180),

Healthy controls are only assessed at Tp1,2,4,5

ELIGIBILITY:
Inclusion Criteria:

ECT:

* Patients (>18) referred to the center of ECT and accepted for treatment
* because of moderate and severe depression
* fulfilling the criteria for the following ICD-10 diagnosis: F 31.3 and F31.4; F32.1 and F32.2 and F32.3; F33.1 and F33.2 and F33.3.
* In addition, the symptom intensity must be verified by a MADRS score ≥ 25.
* There is no upper age for participation, however, the responsible clinician will consider if patients are eligible for inclusion (functioning, enabled to give informed consent).

TMS:

* Patients (>18) referred to the center of TMS and accepted for treatment
* because of moderate and severe depression
* fulfilling the criteria for the following ICD-10 diagnosis: F 31.3 and F31.4; F32.1 and F32.2 and F32.3; F33.1 and F33.2 and F33.3.
* In addition, the symptom intensity must be verified by a MADRS score ≥ 25.
* There is no upper age for participation, however, the responsible clinician will consider if patients are eligible for inclusion (functioning, enabled to give informed consent).

Healthy controls:

* Age and gender matched (to the patient groups).
* No history of psychiatric illness and no current depression.
* No contraindication for MRI scanning.

Exclusion Criteria:

* ECT / TMS treatment within the last 12 months.
* Patients unable to give informed consent (according to the responsible clinician or ECT / TMS responsible).
* Patients who cannot participate in the MR scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients accepted for ECT or TMS at Haukeland University Hospital will be included.
  Control groups: Healthy controls undergoing the same investigations as the ECT and TMS patient groups, but not receiving any treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cerebral Blood Flow from baseline | Baseline, day1 (after 1 ECT), ~ day 15 (after 6 ECTs), ~ day 30 - 50 (1-2 weeks after last ECT), ~ day 180 (6 months after treatment)
  Estimated by Arterial Spin Labeling MRI
Change in MADRS from baseline | Baseline, day1 (after 1 ECT), ~ day 15 (after 6 ECTs), ~ day 30 - 50 (1-2 weeks after last ECT), ~ day 180 (6 months after treatment)
  Depression rating by MADRS score

SECONDARY OUTCOMES:
Change fraction of in Isotropic hindered water | Baseline, day1 (after 1 ECT), ~ day 15 (after 6 ECTs), ~ day 30 - 50 (1-2 weeks after last ECT), ~ day 180 (6 months after treatment)
  Measured by Restriction spectrum imaging. Increase in the fraction of isotropic hindered water as a sign of oedema / disruptive effects of ECT seen on Imaging at 2 hours after first ECT.
Change in concentration of NAA, Choline, myo Inositol | Baseline, day1 (after 1 ECT), ~ day 15 (after 6 ECTs), ~ day 30 - 50 (1-2 weeks after last ECT), ~ day 180 (6 months after treatment)
  MR Spectroscopy og the amygdala, measures of neuronal integrity.
Changes in structural MRI T1 and T2 and RSI | Baseline, day1 (after 1 ECT), ~ day 15 (after 6 ECTs), ~ day 30 - 50 (1-2 weeks after last ECT), ~ day 180 (6 months after treatment)
  Measures of brain structure
Changes in functional MRI | Baseline, day1 (after 1 ECT), ~ day 15 (after 6 ECTs), ~ day 30 - 50 (1-2 weeks after last ECT), ~ day 180 (6 months after treatment)
  Resting state MRI, measurement of functional connectivity
Change in performance on test of spatial navigation | Baseline, day1 (after 1 ECT), ~ day 15 (after 6 ECTs), ~ day 30 - 50 (1-2 weeks after last ECT), ~ day 180 (6 months after treatment)
  Neurocognitive assessments of spatial navigation

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

REFERENCES:
- [Derived] Frid LM, Kessler U, Ousdal OT, Hammar A, Haavik J, Riemer F, Hirnstein M, Ersland L, Erchinger VJ, Ronold EH, Nygaard G, Jakobsen P, Craven AR, Osnes B, Alisauskiene R, Bartsch H, Le Hellard S, Stavrum AK, Oedegaard KJ, Oltedal L. Neurobiological mechanisms of ECT and TMS treatment in depression: study protocol of a multimodal magnetic resonance investigation. BMC Psychiatry. 2023 Oct 30;23(1):791. doi: 10.1186/s12888-023-05239-0. PMID 37904091